CLINICAL TRIAL: NCT07078877
Title: Investigation of Sarcopenia in Patients With Knee Osteoarthritis and the Effect of Low-Level Laser Therapy on Sonographically Measured Femoral Cartilage and Quadriceps Thickness, Clinical Outcomes, and Regional Sarcopenia
Brief Title: Low-Level Laser Therapy in Knee Osteoarthritis: Effects on Clinical Outcomes, Femoral Cartilage Thickness and Regional Sarcopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, IREM ADIGUZEL, Dr, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-058
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Low Level Laser Therapy; Regional Sarcopenia; Exercise Theraphy
Keywords: knee osteoarthritis; low level laser therapy; regional sarcopenia; Exercise Therapy; sarcopenia
MeSH Terms: conditions — Osteoarthritis, Knee; Sarcopenia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Active Comparator): The patients in this group will receive a conventional home-based exercise program.
  Interventions: Other: home based exercise
- exercise and LLLT group (Experimental): This group of patients will receive LLLT treatment in addition to conventional home-based exercise program.
  Interventions: Other: home based exercise; Device: Low Level Laser Therapy

INTERVENTIONS:
Other: home based exercise — The conventional home based exercise program includes: hip and knee range of motion (ROM) exercises; stretching exercises for the hamstring, calf, and quadriceps muscles; isometric, concentric, and eccentric strengthening exercises for the quadriceps, hamstrings, and hip adductors/abductors; relaxation exercises; and walking as aerobic exercises. The program will begin with ROM, stretching, relaxation, aerobic, and isometric strengthening exercises. After one week, concentric and eccentric strengthening exercises will be added using elastic bands. The home exercise program will be performed 3 days a week, each exercise in 3 sets of 10 repetitions and 2 minutes of rest between sets. Aerobic walking at a moderate pace (as determined by the talk test: the patient can talk but not sing during exercise) for 30 minutes will be recommended. Program will continue for 12 weeks.
Device: Low Level Laser Therapy — Patients will receive LLLT treatment, they will be treated in a supine position with the knee flexed to 30 degrees, 5 sessions per week for 2 weeks. A total of 6 points will be treated each for 60 seconds. The treatment will be applied using the BTL SMART 4000 laser device at a wavelength of 835 nm and a dose of 10 J/point.
  Arms: exercise and LLLT group

SUMMARY:
It was designed as a single-center, prospective, randomized controlled study. The study consists of two groups. Both groups of patients will receive a conventional home based exercise program.

In addition to the conventional exercise program, patients in the first group will also receive low-level laser therapy (LLLT). If the laser group is found to be superior at the end of the study, the patients who only received the exercise program will be recalled and administered LLLT. Patients who meet the inclusion criteria will be enrolled in the study.

Sample size calculations were based on data from a previous study by Alghadir et al. Using a mean of 3.25 and a standard deviation of 2.61 for the WOMAC pain subscale, the number of participants was calculated with 95% power and a 5% significance level. As a result, it was determined that at least 29 patients would be included in each group. Written informed consent will be obtained from each patient before enrollment. Randomization will be performed according to the order of patient admissions. Patients will be evaluated before treatment, and at the 1st and 3rd months post-treatment.

The dosage of laser application was selected based on the recommendations of the World Association for Photobiomodulation Therapy (WALT). Patients will be treated 5 sessions per week for 2 weeks. The treatment will be applied using the BTL SMART 4000 laser device at a wavelength of 835 nm and a dose of 10 J/point.

The conventional home based exercise program includes: range of motion (ROM) exercises, stretching, strengthening, relaxation and aerobic exercises. The program will begin with ROM, stretching, relaxation, aerobic, and isometric strengthening exercises. After one week, concentric and eccentric strengthening exercises will be added using elastic bands. The home exercise program will be performed 3 days a week, each exercise in 3 sets of 10 repetitions and 2 minutes of rest between sets. Aerobic walking at a moderate pace for 30 minutes will be recommended. Each patient will be shown and taught the exercises to be performed at home, and will also be provided with illustrated instructions. The home based exercise program will continue for 12 weeks. Patients will be contacted by phone weekly during the first month, and then every two weeks thereafter, to assess their adherence to and continuation of the home based exercise program.

Before starting treatment, demographic information will be collected, medical history will be taken, and a physical examination will be performed. Pre-treatment evaluations include:

* Measurement of height, weight, and calculation of body mass index (BMI)
* Femoral cartilage thickness and quadriceps muscle thickness measurement via ultrasound
* Determination of the Sonographic Thigh Adjustment Ratio (STAR)
* Application of the SARC-F screening test; those scoring over 4 will undergo whole-body muscle mass measurement
* Handgrip strength (HGS) measurement using a Jamar hand dynamometer
* Five-times chair stand test (CST)
* Timed Up and Go (TUG) test
* Six-minute walk test
* Visual Analog Scale (VAS) for pain
* Western Ontario and McMaster Universities Arthritis Index (WOMAC)
* Short Form-36 (SF-36) quality of life questionnaire

Post-treatment evaluations (At the end of the 1st month and at the end of the 3rd month) include:

* Calculation of body mass index (BMI)
* Femoral cartilage thickness and quadriceps muscle thickness (USG)
* STAR index calculation
* Handgrip strength using Jamar dynamometer
* Five-times chair stand test
* Timed Up and Go test
* Six-minute walk test
* Visual Analog Scale (VAS) for pain
* WOMAC
* SF-36 Quality of Life Questionnaire

DETAILED DESCRIPTION:
It was designed as a single-center, prospective, randomized controlled study. The study consists of two groups. Both groups of patients will receive a conventional treatment program. Within the scope of the conventional treatment program, an exercise program (including range of motion, stretching, relaxation, strengthening, and aerobic exercises) will be administered.

In addition to the conventional treatment program, patients in the first group will also receive low-level laser therapy (LLLT). If the laser group is found to be superior at the end of the study, the patients who only received the exercise program will be recalled and administered LLLT. Patients who meet the inclusion criteria will be enrolled in the study.

Sample size calculations were based on data from a previous study by Alghadir et al. Using a mean of 3.25 and a standard deviation of 2.61 for the WOMAC pain subscale, the number of participants was calculated with 95% power and a 5% significance level. As a result, it was determined that at least 29 patients would be included in each group. Written informed consent will be obtained from each patient before enrollment. Randomization will be performed according to the order of patient admissions. Patients will be evaluated before treatment, and at the 1st and 3rd months post-treatment.

The dosage of laser application was selected based on the recommendations of the World Association for Photobiomodulation Therapy (WALT). Patients will be treated 5 sessions per week for 2 weeks. A total of 6 points will be treated, each for 60 seconds. The treatment will be applied using the BTL SMART 4000 laser device at a wavelength of 835 nm and a dose of 10 J/point.

The conventional home based exercise program includes: hip and knee range of motion (ROM) exercises; stretching exercises for the hamstring, calf, and quadriceps muscles; isometric, concentric, and eccentric strengthening exercises for the quadriceps, hamstrings, and hip adductors/abductors; relaxation exercises; and walking as aerobic exercises. The program will begin with ROM, stretching, relaxation, aerobic, and isometric strengthening exercises. After one week, concentric and eccentric strengthening exercises will be added using elastic bands. The home based exercise program will be performed 3 days a week, each exercise in 3 sets of 10 repetitions and 2 minutes of rest between sets. Aerobic walking at a moderate pace (as determined by the talk test: the patient can talk but not sing during exercise) for 30 minutes will be recommended. Each patient will be shown and taught the exercises to be performed at home, and will also be provided with illustrated instructions. The home based exercise program will continue for 12 weeks. Patients will be contacted by phone weekly during the first month, and then every two weeks thereafter, to assess their adherence to and continuation of the home based exercise program.

Before starting treatment, demographic information will be collected, medical history will be taken, and a physical examination will be performed. Pre-treatment evaluations include:

* Measurement of height, weight, and calculation of body mass index (BMI)
* Femoral cartilage thickness and quadriceps muscle thickness measurement via ultrasound
* Determination of the Sonographic Thigh Adjustment Ratio (STAR)
* Application of the SARC-F screening test; those scoring over 4 will undergo whole-body muscle mass measurement
* Handgrip strength (HGS) measurement using a Jamar hand dynamometer
* Five-times chair stand test (CST)
* Timed Up and Go (TUG) test
* Six-minute walk test
* Visual Analog Scale (VAS) for pain
* Western Ontario and McMaster Universities Arthritis Index (WOMAC)
* Short Form-36 (SF-36) quality of life questionnaire

Post-treatment evaluations (At the end of the 1st month and at the end of the 3rd month) include:

* Calculation of body mass index (BMI)
* Femoral cartilage thickness and quadriceps muscle thickness (USG)
* STAR index calculation
* Handgrip strength using Jamar dynamometer
* Five-times chair stand test
* Timed Up and Go test
* Six-minute walk test
* Visual Analog Scale (VAS) for pain
* WOMAC
* SF-36 Quality of Life Questionnaire

ELIGIBILITY:
Inclusion Criteria:

Individuals with knee osteoarthritis according to ACR criteria, Those at grade 2-3 according to the Kellgren-Lawrence scale, Individuals aged over 50 years

Exclusion Criteria:

Individuals with a history of trauma or surgery to the knee joint, Those who have received intra-articular injection to the knee within the last 3 months, Those who have undergone physical therapy or exercise treatment in the past year, Individuals with a pacemaker, Patients with high cardiac risk, Those with active malignancy, Individuals with genetic bone or joint disease, Those with a BMI > 35 kg/m²

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | The scale will be administered to all patients before starting treatment, at the 1st and 3rd months after the initiation of treatment.
  The WOMAC consists of 24 questions divided into 3 subscales. Each question is scored on a scale from 0 to 4, with the scores corresponding to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores are summed for each subscale.

SECONDARY OUTCOMES:
Femoral cartilage thickness | Ultrasound measurements will be performed on all patients during the pre-treatment assessment, as well as at the 1st and 3rd months after treatment.
  The patient will be asked to bring their knee into full flexion while lying in the supine position. Medial, lateral, and intercondylar femoral cartilage thickness will be measured using ultrasound with a 5- to 12-MHz linear probe.
Quadriceps Muscle Thickness | Ultrasound measurements will be performed on all patients during the pre-treatment assessment, as well as at the 1st and 3rd months after treatment.
  The rectus femoris and vastus intermedius of the quadriceps femoris will be evaluated. Measurements will be performed as described in previous studies. While the patient lies in a relaxed supine position, a transverse image will be obtained with ultrasound using linear probe from the midpoint of the line between the anterior superior iliac spine (ASIS) and the superior border of the patella. The average of three measurements of the vastus intermedius and rectus femoris muscles will be recorded as the muscle thickness.
Determination Sonographic Thigh Adjustment Ratio (STAR) value | The STAR value will be measured to all patients before the start of the study, as well as at the 1st and 3rd months after the study begins.
  For the assessment of regional sarcopenia, the Sonographic Thigh Adjustment Ratio (STAR) value will be determined as described in previous studies. Anterior thigh muscle thickness will be measured using ultrasound, and the STAR value will be calculated by dividing the anterior thigh muscle thickness by the body mass index (BMI). In previous studies, STAR cutoff values for diagnosing sarcopenia were identified as 1.0 for women and 1.4 for men.
Visual analog scale pain score | The VAS pain score will be administered to all patients during the pre-treatment assessment, as well as at the 1st and 3rd months after treatment.
  The patient will be shown the VAS pain scale and asked to select their pain level both at rest and during movement. The score will increase as the pain intensifies, and the results will be recorded.
Five times chair stand test (CST) | The test will be administered to all patients before starting treatment, as well as at the 1st and 3rd months after the initiation of treatment.
  The patient is asked to cross their arms in front, stand up and sit down five times. The stopwatch is started as the patient begins to stand up and stopped after completing five repetitions. The duration is recorded in seconds.
Timed Up and Go (TUG) | The test will be administered to all patients before starting treatment, as well as at the 1st and 3rd months after the initiation of treatment.
  The patient crosses their arms in front and stands up without support. The stopwatch is started as the patient begins to stand. The patient walks 3 meters, turns around, and returns to sit down. The stopwatch is stopped once the patient is seated again. The time is recorded in seconds.
Hand Grip Strength | The measurment will be administered to all patients before starting treatment, as well as at the 1st and 3rd months after the initiation of treatment.
  Patients' hand grip strength will be measured using a Jamar hand dynamometer. The measurements will be taken While the patients are seated with their shoulders in adduction and neutral position, elbows flexed at 90 degrees, and forearms/wrists in a neutral position.
6 minutes walk test | The test will be administered to all patients before starting treatment, as well as at the 1st and 3rd months after the initiation of treatment.
  In the 6-minute walk test, the patient is instructed to walk as far as possible without running along a straight corridor of at least 30 meters. At the end of 6 minutes, the total distance walked is measured.
The Short Form 36 (SF-36) | The scale will be administered to all patients before starting treatment, at the 1st and 3rd months after the initiation of treatment.
  The Short Form 36 (SF-36) is a health survey which includes 36 questions. It involves 8 different assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, YENIMAHALLE, Turkey (Türkiye)

REFERENCES:
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Ganjeh S, Rezaeian ZS, Mostamand J. Low Level Laser Therapy in Knee Osteoarthritis: A Narrative Review. Adv Ther. 2020 Aug;37(8):3433-3449. doi: 10.1007/s12325-020-01415-w. Epub 2020 Jul 3. PMID 32621270
- [Background] Chow R, Liebert A, Tilley S, Bennett G, Gabel CP, Laakso L. Guidelines versus evidence: what we can learn from the Australian guideline for low-level laser therapy in knee osteoarthritis? A narrative review. Lasers Med Sci. 2021 Mar;36(2):249-258. doi: 10.1007/s10103-020-03112-0. Epub 2020 Aug 8. PMID 32770424
- [Background] Stausholm MB, Naterstad IF, Joensen J, Lopes-Martins RAB, Saebo H, Lund H, Fersum KV, Bjordal JM. Efficacy of low-level laser therapy on pain and disability in knee osteoarthritis: systematic review and meta-analysis of randomised placebo-controlled trials. BMJ Open. 2019 Oct 28;9(10):e031142. doi: 10.1136/bmjopen-2019-031142. PMID 31662383
- [Background] Bennell KL, Hinman RS. A review of the clinical evidence for exercise in osteoarthritis of the hip and knee. J Sci Med Sport. 2011 Jan;14(1):4-9. doi: 10.1016/j.jsams.2010.08.002. Epub 2010 Sep 17. PMID 20851051
- [Background] Raposo F, Ramos M, Lucia Cruz A. Effects of exercise on knee osteoarthritis: A systematic review. Musculoskeletal Care. 2021 Dec;19(4):399-435. doi: 10.1002/msc.1538. Epub 2021 Mar 5. PMID 33666347
- [Background] Alghadir A, Omar MT, Al-Askar AB, Al-Muteri NK. Effect of low-level laser therapy in patients with chronic knee osteoarthritis: a single-blinded randomized clinical study. Lasers Med Sci. 2014 Mar;29(2):749-55. doi: 10.1007/s10103-013-1393-3. Epub 2013 Aug 3. PMID 23912778
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Background] Kholvadia A, Constantinou D, Gradidge PJ. Exploring the efficacy of low-level laser therapy and exercise for knee osteoarthritis. S Afr J Sports Med. 2019 Jan 1;31(1):v31i1a6058. doi: 10.17159/2078-516X/2019/v31i1a6058. eCollection 2019. PMID 36817986
- See also: World Association of Laser Therapy — https://waltpbm.org/wp-content/uploads/2021/08/Dose_table_780-860nm_for_Low_Level_Laser_Therapy_WALT-2010.pdf